CLINICAL TRIAL: NCT07229651
Title: Safety and Efficacy of Metformin in Patients With Parkinson Disaese
Brief Title: Metformin in Parkinson Disease
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ihab Elsayed Hassan, Lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4258
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Double blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Control group (Levo-dopa group, n =30) who will receive levodopa/carbidopa (125/12.5 mg) three times daily for 6 months
  Interventions: Drug: Levodopa Carbidopa
- Metformin group (Active Comparator): Patients will receive levodopa/carbidopa (125/12.5 mg) three times daily plus metformin 500 mg two times daily for 6 months
  Interventions: Drug: Levodopa Carbidopa; Drug: Metformin

INTERVENTIONS:
Drug: Levodopa Carbidopa — Carbidopa/levodopa, also known as levocarb and co-careldopa, is the combination of the two medications carbidopa and levodopa. It is primarily used to manage the symptoms of Parkinson's disease
Drug: Metformin — Metformin, sold under the brand name Glucophage, among others, is the main first-line medication for the treatment of type 2 diabetes, particularly in people who are overweight.
  Arms: Metformin group

SUMMARY:
The clinical manifestations of Parkinson's disease (PD), a chronic neurodegenerative condition, include resting tremor, hypokinesia, bradykinesia, stiffness and postural instability. These motor symptoms are caused by a selective loss and degeneration of dopaminergic neurons in the substantia nigra pars compacta (SNpc) region, which leads to a dopamine (DA) insufficiency in the striatum

ELIGIBILITY:
Inclusion Criteria:

Eligible participants were men and women aged 50 years or older with a confirmed diagnosis of PD Patients receiving levodopa/carbidopa therapy.

Exclusion Criteria:

Secondary causes of parkinsonism Patients taking anti-inflammatory drugs Atypical parkinsonian syndromes Prior stereotaxic surgery for Parkinson's disease Pregnancy and lactation Cardiovascular disease patients Patients with coagulation disorders Suffering from active malignancy Addiction to alcohol and / or drugs Known allergy to the studied medications

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-11-20 (Estimated); Study Completion 2027-09-20 (Estimated)

PRIMARY OUTCOMES:
change in The Unified Parkinson's Disease Rating Scale (UPDRS). | 6 months
  The unified Parkinson's disease rating scale is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease.

SECONDARY OUTCOMES:
Change in PDQ-39 | 6 months
  The Parkinson's Disease Questionnaire-39 (PDQ-39) is a widely recognized, disease-targeted, self-administered tool that captures patients' perspectives on how Parkinson's disease influences their health-related quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt